CLINICAL TRIAL: NCT06507488
Title: Daphnetin Capsule In the Treatment of VaScular COgnitive Impairment Without Dementia - A Randomized, Double-blind, Placebo-controlled Study
Brief Title: Daphnetin Capsule In the Treatment of VaScular COgnitive Impairment Without Dementia
Acronym: DISCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Shenyang (Other)
Collaborators: The Fourth People's Hospital of Shenyang (Unknown)
Responsible Party: Principal Investigator, Dr. Yi Sui, vice president, Fourth People's Hospital of Shenyang
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RXSJNJLXD-2024-SYSY
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Cerebrovascular Disorders
Keywords: Vascular Cognitive Impairment No Dementia; Daphnetin; Effectiveness; safety
MeSH Terms: conditions — Cerebrovascular Disorders | interventions — daphnetin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daphnetin (Experimental): oral Daphnetin Capsule three capsules/tid for up to six months.
  Interventions: Drug: Daphnetin Capsule
- Placebo (Placebo Comparator): oral Placebo (Daphnetin Capsule simulants) three capsules/tid for up to six months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Daphnetin Capsule — Daphnetin, chemically known as 7,8-dihydroxycoumarin, also known as ZuShiMaJiaSu, is a class of coumarin derivatives derived from different Daphnetin genus plant .
  Other Names: 7,8-dihydroxycoumarin
  Arms: Daphnetin
Drug: Placebo — The placebo is a Daphnetin Capsule simulants
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to understand and evaluate the clinical efficacy and safety of Daphnetin Capsule in patients with vascular cognitive impairment. Changes in the Vascular Dementia Assessment Scale-cog(VADAS-cog) at 6 months were evaluated. Although Daphnetin has a dual neurovascular protective effect, however, there is still a lack of relevant high-quality studies on its role in patients with vascular cognitive impairment, especially in patients with vascular cognitive impairment in non-dementia (VCI-ND), whether it has a role in improving cognitive status needs to be urgently explored in high-quality clinical studies. Researchers are comparing Daphnetin to placebo (a drug-free analog) to see if Daphnetin is effective in treating vascular cognitive impairment. Participants will take either Daphnetin or placebo daily for six months, with follow-up visits every three months and completion of a case report form.

DETAILED DESCRIPTION:
Vascular cognitive impairment (VCI) is caused by ischemic or hemorrhagic strokes and other cerebrovascular diseases, leading to cognitive and memory function impairment. With the aging population and high incidence of cerebrovascular diseases in China, Vascular cognitive impairment (VCI) prevalence is rising, increasing the disease burden. However, due to the complexity of Vascular cognitive impairment (VCI) symptoms and imaging changes, targeted therapies are currently lacking.

Daphnetin, a coumarin derivative, has shown promise in treating various diseases and has gained significant attention recently. It offers "triple protection" for blood, blood vessels, and ischemic tissues by inhibiting inflammation, anticoagulation, and thrombosis, protecting endothelial structures, and regulating vasoactive substances. Daphnetin is particularly beneficial for cardio-cerebral vascular disease, diabetes mellitus, and microvascular complications. It also expands peripheral blood vessels, improving circulation and alleviating vascular occlusive diseases.

Research indicates that Daphnetin's anti-inflammatory effects can inhibit neuroinflammation, promote synaptic growth, and enhance neuronal survival, protecting nerve cells and repairing damage. Despite these benefits, there is a lack of high-quality studies on Daphnetin's role in non-dementia vascular cognitive impairment (VCI-ND).

This project aims to evaluate the clinical efficacy and safety of oral Daphnetin capsules in treating Vascular cognitive impairment (VCI) through a prospective, randomized, double-blind, placebo-controlled study. Patients with vascular cognitive dysfunction confirmed by cerebral small vessel disease imaging will participate. The study will follow the international FINESSE framework, comparing Daphnetin to a placebo over six months, with follow-up visits and case report forms completed every three months.

ELIGIBILITY:
Inclusion Criteria:

1. Be 50-80 years of age (both ends included)
2. Have a complaint of cognitive impairment involving memory and/or other cognitive domains that has persisted for at least 3 months
3. Have a cognitive level that is neither normal nor demented according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Criteria ( DSM-V criteria）, a Montreal Cognitive Assessment (MoCA scale) score <26 and ≥18, and a Clinical Dementia Rating (CDR) scale score of ≥0.5 in at least one domain and an overall CDR score ≤1
4. Have a cognitive level that is neither normal nor demented according to DSM-V criteria, a MoCA scale score <26 and ≥18, and a CDR scale score of ≥0.5 in at least one domain and an overall CDR score ≤1
5. Voluntarily participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Previously diagnosed dementia; vascular cognitive impairment not associated with a condition other than dementia that may affect cognition
2. Acute stroke event within 6 months
3. Previously diagnosed hereditary or inflammatory small vessel disease
4. Presence of congenital mental retardation and severe neurological or psychiatric disorders
5. Illiteracy or severe visual or hearing impairment, severe aphasia, and other factors that may preclude cooperation with neuropsychological evaluation
6. Associated depression (Hamilton Depression Scale score ≥ 17), or other unrelated serious mental illness (schizophrenia, bipolar disorder, or delirium)
7. Combined severe cardiac, pulmonary, and renal insufficiency (creatinine > 2.0 mg/dl or 177 μ mol/L), and severe hepatic impairment (aminotransferases more than 3 times normal)
8. Alcoholism, drug addiction, or ongoing use of medications that affect cognitive assessment, such as tranquilizers, sleeping pills, puberty pills, and cholinergics
9. Malignant tumors that have been clearly diagnosed, vital organ failure
10. Those with bleeding tendency after surgery
11. Pregnant and lactating women are prohibited
12. Severe hypertension (Systolic Blood Pressure(SBP)≥160mmHg and/or Diastolic Blood Pressure(DBP)≥110mmHg) is prohibited
13. Previous allergy or intolerance to the ingredients of Reserpine
14. The subject does not have a stable and reliable caregiver or the caregiver is unable to assist the subject in participating in the study
15. Patients who have participated in other interventional clinical studies within the last 3 months or are currently participating in other interventional clinical studies.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Vascular Dementia Assessment Scale-cognitive subscale (VADAS-cog) | 6 months
  Vascular Dementia Assessment Scale-cognitive subscale（VADAS-cog） is a revision of the Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-cog) to be a better measure in vascular conditions，The lowest score is 0, with higher scores representing higher levels of cognitive dysfunction and poorer status of the patient.

SECONDARY OUTCOMES:
Incidence of combined endpoints: including new stroke (ischemic Trial of ORG 10172 in Acute Stroke Treatment typing [TOAST typing] or hemorrhagic)/transient ischemic attack, myocardial infarction, new-onset dementia, death | 6 months
  For categorical indicators, the stratified Cochran- Mantel-Haenszel (CMH) test will be used for analysis.
Incidence of each individual event of the combined endpoint | 6 months
  For categorical indicators, the stratified Cochran- Mantel-Haenszel (CMH) test will be used for analysis.
Clinician Interview-Based studies Impression of Change scale-plus version(CIBIC-Plus) of change | 6 months
  Consists of three parts The clinician's impression of change is an assessment of change from baseline, not an assessment of severity. The clinician may refer to his/her own baseline information compiled in Part I when making the assessment of change. The clinician's assessment of impression of change should then be replicated in the main study case report form.The score of CIBIC-plus ranges from 1 to 7, and the score of 1-3 indicates improvement, 4 means no changed, and 5-7 indicates worse.
Change in the Brief Mental State Evaluation Scale (MMSE) | 6 months
  Each correct item is scored as 1 point, and errors are scored as 0 points. The total score ranges from 0 to 30, and the cut-off value for normal and abnormal is related to the level of education; ≤17 points for the illiterate (no education) group, ≤20 points for the elementary school (≤6 years of education) group, and ≤24 points for the secondary school or above (>6 years of education) group. Cognitive deficits are considered to be below the cut-off value and normal above it.
Change in the Montreal Cognitive Assessment Scale (MoCA) | 6 months
  The MoCA scale is a 30-point scale, with ≥26 normal, 18-26 mild cognitive impairment (MCI), 10-17 moderate, and less than 10 severe.Patients with MCI scored approximately 22 (19-25) points, and patients with AD scored between 11-21 points.
Changes in the Symbol Digit Transformation Test (SDMT) | 6 months
  Completion of the SDMT scale within 90 seconds, with a total score of 0-110; the lower the score, the more severe the degree of cognitive impairment
Change in Clinical Dementia Rating Scale (CDR) | 6 months
  The total score ranges from 0 to 18,The higher the score, the more demented the patient is, the worse the state is.
Change in Neuropsychiatric Questionnaire (NPI-Q) | 6 months
  Presence of symptoms (1-2): 1=present 2=absent. Frequency (1-4 points): 1=occasional, less than weekly; 2=frequent, about weekly; 3=several times a week but less than daily; 4=very frequent, once or more at a time or continuously.
  Severity (on a scale of 1 to 3): 1=mild, perceptible but not obvious; 2=moderate, obvious but not very prominent; 3=severe, very prominent changes.
  The degree of distress caused by the symptom to the caregiver (0-5 points): 0 = no distress; 1 = very mild distress, caregiver does not need to take steps to cope; 2 = mild distress, caregiver copes easily; 3 = moderate distress, caregiver struggles to cope; 4 = severe, caregiver is barely able to cope; 5 = extreme distress, caregiver is unable to cope. The higher the score the more severe
Changes in the Activities of Daily Living Scale (ADL) | 6 months
  1 = can do it all by myself; 2 = can still do it with some difficulty; 3 = need help 4 = cannot do it at all. When the patient never does it but is able to do it, it is rated as 1, never does it but has difficulty doing it but does not need help, 2, never does it but needs help, 3, never does it and is unable to do it, 4. The range of scores is from 20 to 80, and a score of >23 is considered to be cognitively impaired.
Changes in motor function (TUG, time to walk three meters) | 6 months
  Change in motor score (TUG, time to walk three meters) at 6 months relative to baseline
EuroQol Five Dimensions Questionnaire (EQ-5D) | 6 months
  The EuroQol Five Dimensions Questionnaire (EQ-5D) health description system consists of five dimensions: mobility (MO), self-care (SC), ability to perform activities of daily living (UA), pain or discomfort (PD), and anxiety or depression (AD), each of which can be reported separately as "no problem, moderate problem, or severe problem".Self-rated health on a scale of 0 to 100, the higher the score the better your health is considered to be.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Sui, MD PhD, Principal Investigator — The Fourth People's Hospital of Shenyang, China Medical University
Locations (1):
- Shenyang First People's Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Benisty S. [Current concepts in vascular dementia]. Geriatr Psychol Neuropsychiatr Vieil. 2013 Jun;11(2):171-80. doi: 10.1684/pnv.2013.0410. French. PMID 23803634
- [Background] Wu YT, Lee HY, Norton S, Chen C, Chen H, He C, Fleming J, Matthews FE, Brayne C. Prevalence studies of dementia in mainland china, Hong Kong and taiwan: a systematic review and meta-analysis. PLoS One. 2013 Jun 11;8(6):e66252. doi: 10.1371/journal.pone.0066252. Print 2013. PMID 23776645
- [Background] D'Onofrio G, Sancarlo D, Addante F, Ciccone F, Cascavilla L, Paris F, Picoco M, Nuzzaci C, Elia AC, Greco A, Chiarini R, Panza F, Pilotto A. Caregiver burden characterization in patients with Alzheimer's disease or vascular dementia. Int J Geriatr Psychiatry. 2015 Sep;30(9):891-9. doi: 10.1002/gps.4232. Epub 2014 Dec 4. PMID 25475248
- [Background] Kalaria RN. The pathology and pathophysiology of vascular dementia. Neuropharmacology. 2018 May 15;134(Pt B):226-239. doi: 10.1016/j.neuropharm.2017.12.030. Epub 2017 Dec 19. PMID 29273521
- [Background] Plassman BL, Langa KM, Fisher GG, Heeringa SG, Weir DR, Ofstedal MB, Burke JR, Hurd MD, Potter GG, Rodgers WL, Steffens DC, Willis RJ, Wallace RB. Prevalence of dementia in the United States: the aging, demographics, and memory study. Neuroepidemiology. 2007;29(1-2):125-32. doi: 10.1159/000109998. Epub 2007 Oct 29. PMID 17975326
- [Background] Javed M, Saleem A, Xaveria A, Akhtar MF. Daphnetin: A bioactive natural coumarin with diverse therapeutic potentials. Front Pharmacol. 2022 Sep 29;13:993562. doi: 10.3389/fphar.2022.993562. eCollection 2022. PMID 36249766
- [Background] Singh L, Singh AP, Bhatti R. Mechanistic interplay of various mediators involved in mediating the neuroprotective effect of daphnetin. Pharmacol Rep. 2021 Oct;73(5):1220-1229. doi: 10.1007/s43440-021-00261-z. Epub 2021 Apr 16. PMID 33860917
- [Background] Chaudhary PK, Kim S, Kim S. Antiplatelet Effect of Daphnetin Is Regulated by cPLA2-Mediated Thromboxane A2 Generation in Mice. Int J Mol Sci. 2023 Mar 17;24(6):5779. doi: 10.3390/ijms24065779. PMID 36982853
- [Background] Syed AM, Kundu S, Ram C, Kulhari U, Kumar A, Mugale MN, Mohapatra P, Murty US, Sahu BD. Up-regulation of Nrf2/HO-1 and inhibition of TGF-beta1/Smad2/3 signaling axis by daphnetin alleviates transverse aortic constriction-induced cardiac remodeling in mice. Free Radic Biol Med. 2022 Jun;186:17-30. doi: 10.1016/j.freeradbiomed.2022.04.019. Epub 2022 May 2. PMID 35513128
- [Background] Yang F, Jiang X, Cao H, Shuai W, Zhang L, Wang G, Quan D, Jiang X. Daphnetin Preconditioning Decreases Cardiac Injury and Susceptibility to Ventricular Arrhythmia following Ischaemia-Reperfusion through the TLR4/MyD88/NF-Kappab Signalling Pathway. Pharmacology. 2021;106(7-8):369-383. doi: 10.1159/000513631. Epub 2021 Apr 26. PMID 33902056
- [Background] Yang Y, Sheng Q, Nie Z, Liu L, Zhang W, Chen G, Ye F, Shi L, Lv Z, Xie J, Wang D. Daphnetin inhibits spinal glial activation via Nrf2/HO-1/NF-kappaB signaling pathway and attenuates CFA-induced inflammatory pain. Int Immunopharmacol. 2021 Sep;98:107882. doi: 10.1016/j.intimp.2021.107882. Epub 2021 Jun 26. PMID 34182245
- [Background] Du G, Tu H, Li X, Pei A, Chen J, Miao Z, Li J, Wang C, Xie H, Xu X, Zhao H. Daphnetin, a natural coumarin derivative, provides the neuroprotection against glutamate-induced toxicity in HT22 cells and ischemic brain injury. Neurochem Res. 2014 Feb;39(2):269-75. doi: 10.1007/s11064-013-1218-6. Epub 2013 Dec 17. PMID 24343531
- [Background] Yu W, Wang H, Ying H, Yu Y, Chen D, Ge W, Shi L. Daphnetin attenuates microglial activation and proinflammatory factor production via multiple signaling pathways. Int Immunopharmacol. 2014 Jul;21(1):1-9. doi: 10.1016/j.intimp.2014.04.005. Epub 2014 Apr 18. PMID 24747094
- [Background] Zhi J, Duan B, Pei J, Wu S, Wei J. Daphnetin protects hippocampal neurons from oxygen-glucose deprivation-induced injury. J Cell Biochem. 2019 Mar;120(3):4132-4139. doi: 10.1002/jcb.27698. Epub 2018 Sep 27. PMID 30260007
- [Background] Wang D, Zhu B, Liu X, Han Q, Ge W, Zhang W, Lu Y, Wu Q, Shi L. Daphnetin Ameliorates Experimental Autoimmune Encephalomyelitis Through Regulating Heme Oxygenase-1. Neurochem Res. 2020 Apr;45(4):872-881. doi: 10.1007/s11064-020-02960-0. Epub 2020 Jan 16. PMID 31950453
- [Background] Yang L, Yang Q, Zhang K, Li YJ, Wu YM, Liu SB, Zheng LH, Zhao MG. Neuroprotective effects of daphnetin against NMDA receptor-mediated excitotoxicity. Molecules. 2014 Sep 15;19(9):14542-55. doi: 10.3390/molecules190914542. PMID 25225718
- [Background] Yan L, Zhou X, Zhou X, Zhang Z, Luo HM. Neurotrophic effects of 7,8-dihydroxycoumarin in primary cultured rat cortical neurons. Neurosci Bull. 2012 Oct;28(5):493-8. doi: 10.1007/s12264-012-1233-7. Epub 2012 May 18. PMID 22961470
- [Background] Benjamin P, Zeestraten E, Lambert C, Ster IC, Williams OA, Lawrence AJ, Patel B, MacKinnon AD, Barrick TR, Markus HS. Progression of MRI markers in cerebral small vessel disease: Sample size considerations for clinical trials. J Cereb Blood Flow Metab. 2016 Jan;36(1):228-40. doi: 10.1038/jcbfm.2015.113. PMID 26036939
- [Background] Markus HS, van Der Flier WM, Smith EE, Bath P, Biessels GJ, Briceno E, Brodtman A, Chabriat H, Chen C, de Leeuw FE, Egle M, Ganesh A, Georgakis MK, Gottesman RF, Kwon S, Launer L, Mok V, O'Brien J, Ottenhoff L, Pendlebury S, Richard E, Sachdev P, Schmidt R, Springer M, Tiedt S, Wardlaw JM, Verdelho A, Webb A, Werring D, Duering M, Levine D, Dichgans M. Framework for Clinical Trials in Cerebral Small Vessel Disease (FINESSE): A Review. JAMA Neurol. 2022 Nov 1;79(11):1187-1198. doi: 10.1001/jamaneurol.2022.2262. PMID 35969390
- [Background] Pendlebury ST, Mariz J, Bull L, Mehta Z, Rothwell PM. MoCA, ACE-R, and MMSE versus the National Institute of Neurological Disorders and Stroke-Canadian Stroke Network Vascular Cognitive Impairment Harmonization Standards Neuropsychological Battery after TIA and stroke. Stroke. 2012 Feb;43(2):464-9. doi: 10.1161/STROKEAHA.111.633586. Epub 2011 Dec 8. PMID 22156700
- [Background] Ghafar MZAA, Miptah HN, O'Caoimh R. Cognitive screening instruments to identify vascular cognitive impairment: A systematic review. Int J Geriatr Psychiatry. 2019 Aug;34(8):1114-1127. doi: 10.1002/gps.5136. Epub 2019 May 16. PMID 31050033
- [Background] Smith EE, Biessels GJ, De Guio F, de Leeuw FE, Duchesne S, During M, Frayne R, Ikram MA, Jouvent E, MacIntosh BJ, Thrippleton MJ, Vernooij MW, Adams H, Backes WH, Ballerini L, Black SE, Chen C, Corriveau R, DeCarli C, Greenberg SM, Gurol ME, Ingrisch M, Job D, Lam BYK, Launer LJ, Linn J, McCreary CR, Mok VCT, Pantoni L, Pike GB, Ramirez J, Reijmer YD, Romero JR, Ropele S, Rost NS, Sachdev PS, Scott CJM, Seshadri S, Sharma M, Sourbron S, Steketee RME, Swartz RH, van Oostenbrugge R, van Osch M, van Rooden S, Viswanathan A, Werring D, Dichgans M, Wardlaw JM. Harmonizing brain magnetic resonance imaging methods for vascular contributions to neurodegeneration. Alzheimers Dement (Amst). 2019 Feb 26;11:191-204. doi: 10.1016/j.dadm.2019.01.002. eCollection 2019 Dec. PMID 30859119
- [Background] Shi J, Wei M, Ni J, Sun F, Sun L, Wang J, Yu T, Wang K, Lv P, Wang Y, Zhang Y, Gao X, Gao X, Luo B, Mao S, Zhang B, Ren X, Yu F, Hu W, Yin P, Wu N, Liu X, Bi Q, Wang Y, Tian J; CHASE Study Group. Tianzhi granule improves cognition and BPSD of vascular dementia: a randomized controlled trial. J Transl Med. 2020 Feb 13;18(1):76. doi: 10.1186/s12967-020-02232-z. PMID 32054507
- [Background] Smith EE. Clinical presentations and epidemiology of vascular dementia. Clin Sci (Lond). 2017 Jun 1;131(11):1059-1068. doi: 10.1042/CS20160607. PMID 28515342